CLINICAL TRIAL: NCT01083134
Title: The Correlation of Heart Hemodynamic Status Between 320 Multidetector Computed Tomography, Echocardiography and Cardiac Catheterization in Patients With Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 98-4077B
Record Dates: First submitted 2010-03-07; First posted 2010-03-09 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Artery Disease
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- percentage of stenosis

SUMMARY:
With the advances in multidetector computed tomography (MDCT) technology, CT angiography (CTA) of the coronary arteries using 64-slice or dual-source CT systems has evolved into a robust, alternative, noninvasive imaging technique to rule out coronary artery disease (CAD). Reported sensitivities and specificities of coronary CTA can compete with those of catheter angiography.

Because CT is the major source of ionizing radiation in medicine, dual isotope myocardial perfusion scintigraphy and coronary CTA 16-, 64-slice MDCT and DSCT scanners are associated with the highest amount of radiation dose. Recently, a new generation of MDCT machines with even more detector row (320) has become clinically available. The maximum detector width of 16 cm enables the entire heart to be examined in a single rotation and within a single heartbeat and is expected to substantially reduce artifacts from breathing and body motion. Due to high volume coverage, 320-slice CT machines are able to perform a nonspiral, ECG-gated examination of the heart within a single breath-hold.

The purpose of this study was to investigate the correlation of hemodynamic status of 320 MDCT, echocardiography, and coronary catheterization in patients who suspected coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Intermediate or high risk for coronary artery disease
2. Healthy volunteers

Exclusion Criteria:

1. Unstable angina
2. Acute myocardial infarction
3. Active cancer status
4. Renal failure(Creatinine > 1.5 mg/dl)
5. Contrast allergy history
6. Pregnancy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to Diamond and Forrester colleague, there are risks including age, gender, smoking, diabetes, and dyslipidemia for coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Gung Memorial Hospital at Linkou, Taipei, Taiwan

REFERENCES:
- [Background] Achenbach S, Ropers D, Kuettner A, Flohr T, Ohnesorge B, Bruder H, Theessen H, Karakaya M, Daniel WG, Bautz W, Kalender WA, Anders K. Contrast-enhanced coronary artery visualization by dual-source computed tomography--initial experience. Eur J Radiol. 2006 Mar;57(3):331-5. doi: 10.1016/j.ejrad.2005.12.017. Epub 2006 Jan 19. PMID 16426789
- [Background] Hoffmann U, Nagurney JT, Moselewski F, Pena A, Ferencik M, Chae CU, Cury RC, Butler J, Abbara S, Brown DF, Manini A, Nichols JH, Achenbach S, Brady TJ. Coronary multidetector computed tomography in the assessment of patients with acute chest pain. Circulation. 2006 Nov 21;114(21):2251-60. doi: 10.1161/CIRCULATIONAHA.106.634808. Epub 2006 Oct 30. PMID 17075011
- [Background] Johnson TR, Nikolaou K, Wintersperger BJ, Knez A, Boekstegers P, Reiser MF, Becker CR. ECG-gated 64-MDCT angiography in the differential diagnosis of acute chest pain. AJR Am J Roentgenol. 2007 Jan;188(1):76-82. doi: 10.2214/AJR.05.1153. PMID 17179348
- [Background] Scheffel H, Alkadhi H, Plass A, Vachenauer R, Desbiolles L, Gaemperli O, Schepis T, Frauenfelder T, Schertler T, Husmann L, Grunenfelder J, Genoni M, Kaufmann PA, Marincek B, Leschka S. Accuracy of dual-source CT coronary angiography: First experience in a high pre-test probability population without heart rate control. Eur Radiol. 2006 Dec;16(12):2739-47. doi: 10.1007/s00330-006-0474-0. Epub 2006 Sep 19. PMID 17031451
- [Background] Einstein AJ. Radiation risk from coronary artery disease imaging: how do different diagnostic tests compare? Heart. 2008 Dec;94(12):1519-21. doi: 10.1136/hrt.2007.135731. No abstract available. PMID 19011135
- [Background] Hausleiter J, Meyer T, Hadamitzky M, Huber E, Zankl M, Martinoff S, Kastrati A, Schomig A. Radiation dose estimates from cardiac multislice computed tomography in daily practice: impact of different scanning protocols on effective dose estimates. Circulation. 2006 Mar 14;113(10):1305-10. doi: 10.1161/CIRCULATIONAHA.105.602490. Epub 2006 Mar 6. PMID 16520411
- [Background] Yates SJ, Pike LC, Goldstone KE. Effect of multislice scanners on patient dose from routine CT examinations in East Anglia. Br J Radiol. 2004 Jun;77(918):472-8. doi: 10.1259/bjr/21927258. PMID 15151967
- [Background] Hein PA, Romano VC, Lembcke A, May J, Rogalla P. Initial experience with a chest pain protocol using 320-slice volume MDCT. Eur Radiol. 2009 May;19(5):1148-55. doi: 10.1007/s00330-008-1255-8. Epub 2009 Jan 10. PMID 19137311
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Diamond GA, Forrester JS. Analysis of probability as an aid in the clinical diagnosis of coronary-artery disease. N Engl J Med. 1979 Jun 14;300(24):1350-8. doi: 10.1056/NEJM197906143002402. PMID 440357